CLINICAL TRIAL: NCT05117749
Title: The Effect of Saffron in Patients With Ulcerative Colitis: A Randomized Double-blind Clinical Trial
Brief Title: Saffron and Ulcerative Colitis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shiraz University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Ali Reza Safarpour, Manager in chief of gastroenterohepatology research center, Assistant Professor, Shiraz University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 24540
Record Dates: First submitted 2021-10-21; First posted 2021-11-11 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2022-05

CONDITIONS: Ulcerative Colitis
Keywords: saffron; Ulcerative Colitis; inflammatory bowel disease; randomized double-blind clinical trial
MeSH Terms: conditions — Colitis, Ulcerative; Inflammatory Bowel Diseases

STUDY DESIGN:
Intervention Model Description: Sixty eligible patients will be recruited and randomized into 6 groups to receive either saffron capsule or placebo.
Who Masked: Participant, Investigator
Masking Description: Both patients and investigators do not know whether the participant receiving a placebo or saffron.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Mild UC-Saffron 100 (Experimental): Mild UC patients, receiving 100 milligram (mg)/day saffron for 8 weeks (50 mg two times (BID)), n=10
  Interventions: Drug: Saffron 100
- Moderate UC-Saffron 100 (Experimental): Moderate UC patients, receiving100 mg/day saffron for 8 weeks (50 mg BID), n=10
  Interventions: Drug: Saffron 100
- Mild UC-Saffron 50 (Experimental): Mild UC patients, receiving 50 mg/day saffron for 8 weeks (25 mg BID), n=10
  Interventions: Drug: Saffron 50
- Moderate UC-Saffron 50 (Experimental): Moderate UC patients, receiving 50 mg/day saffron for 8 weeks (25 mg BID), n=10
  Interventions: Drug: Saffron 50
- Mild UC-placebo (Placebo Comparator): Mild UC patients, receiving 2 tablets of placebo for 8 weeks, n=10
  Interventions: Drug: Placebo
- Moderate UC-placebo (Placebo Comparator): Moderate UC patients, receiving 2 tablets of placebo for 8 weeks, n=10
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Saffron 100 — to Mild and Moderate UC patients
  Arms: Mild UC-Saffron 100; Moderate UC-Saffron 100
Drug: Saffron 50 — to Mild and Moderate UC patients
  Arms: Mild UC-Saffron 50; Moderate UC-Saffron 50
Drug: Placebo — to Mild and Moderate UC patients
  Arms: Mild UC-placebo; Moderate UC-placebo

SUMMARY:
IBD is a chronic disease with two major types of Crohn's Disease (CD) and Ulcerative Colitis (UC). Nowadays, synthetic drugs and monoclonal antibodies are the most common types of drugs used for IBD management. However, due to their side effects and the high relapse rate, many researchers are looking for plant-derived products to manage the disease. Saffron, Crocus sativus L., is widely used as spice and medicine with anti-obesity, anticonvulsant, anti-hyperlipidemic, anti-tumor, antioxidant, and anti-inflammatory properties. Besides, there is evidence of the favorable effects of saffron on the gut microbiome. The main aim of this proposal is to evaluate the effect of saffron as a complementary supplement or add-on therapy in combination with current therapeutic agents in patients with mild and moderate UC.

DETAILED DESCRIPTION:
This study will be a parallel, randomized, double-blinded clinical trial assessing the efficacy of the saffron extract compared to placebo in patients with mild and moderate UC. Sixty eligible patients will be recruited and randomized into 6 groups to receive either saffron capsule or placebo. Randomization will be performed by an independent researcher (AAK) who is not directly involved in the trial and using software-generated random permuted blocks. Allocation concealment will be also conducted using sealed, opaque envelopes with consecutive numbering. The saffron and placebo will be provided free of charge by Sina Pajoohan Salamat co, Mashhad, Iran. The standard treatment will be administered to all patients as recommendations of the physicians.

Intervention

The intervention groups of study will be included:

1. Mild UC patients, receiving100 milligram (mg)/day saffron for 8 weeks (50 mg two times (BID)), n=10
2. Moderate UC patients, receiving100 mg/day saffron for 8 weeks (50 mg BID), n=10
3. Mild UC patients, receiving 50 mg/day saffron for 8 weeks (25 mg BID), n=10
4. Moderate UC patients, receiving 50 mg/day saffron for 8 weeks (25 mg BID), n=10
5. Mild UC patients, receiving 2 tablets of placebo for 8 weeks, n=10
6. Moderate UC patients, receiving 2 tablets of placebo for 8 weeks, n=10

Demographic and baseline characteristics will be recorded, and assessment of anthropometric and biochemical parameters, fecal calprotectin, inflammatory cytokines, stool microbiome, and its transcriptomic, and metabolomic, urine and saliva metabolomics, health-related quality of life (HRQoL), anxiety, and disease severity will be done at baseline and after 8 weeks. Fecal calprotectin, C-reactive protein (CRP), erythrocyte sedimentation rate (ESR), and disease severity will also be evaluated at 4th week. Moreover, HRQoL and anxiety will also be examined after 6 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients between 18-80 years' old
2. Patients who have received a diagnosis of UC at least 3 months prior to screening. The diagnosis of UC must be confirmed by endoscopic and histologic evidence.
3. Patients with the ability to give written informed consent and to be compliant with the schedule of intervention and assessments
4. Patients with mild (3-5) or moderate (6-11) UC, according to the Simple Clinical Colitis Activity Index

Exclusion Criteria:

1. Pregnant patients or those planning pregnancy
2. Patients receiving immunosuppressive agents for diseases other than UC
3. Patients with confirmed cancer, dysplasia, autoimmune, and rheumatology diseases
4. Patients who had surgery for UC treatment
5. Individuals with liver disease or abnormal liver enzymes and function tests (e.g. total bilirubin, aspartate aminotransferase (AST) or alanine aminotransferase (ALT)) at the screening visit
6. Patients who have any condition affecting oral drug absorption.
7. Subjects with known active or untreated GI infections including C.diff, CMV, HSV, HIV
8. Subjects with clinical features of CD; history of CD (Crohns colitis, or Ileo-colitis), clinical signs of fulminant colitis, toxic megacolon, or Microscopic Colitis, indeterminate Colitis, infectious Colitis, or ischemic colitis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-05 (Estimated); Primary Completion 2025-02 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Changes in clinical response | 4 and 8 weeks
  Changes in clinical response will be assessed by "Simple Clinical Colitis Activity Index", which has a total score between 0 to 19. Higher scores are interpreted to higher disease activity (worse outcome).
Changes in the fecal calprotectin level | 4 and 8 weeks
Changes in the serum levels of CRP | 4 and 8 weeks
Changes in the serum levels of ESR | 4 and 8 weeks

SECONDARY OUTCOMES:
Changes in the serum anti-inflammatory and pro-inflammatory markers | 8 week
  IL-1, IL-6, IL-10, IL-13RA2, IL18, IL17, TREM1, TNF- α, TNFR2, and oncostatin M (pg/ml)
Changes in the Health-related quality of life (HRQoL ) | 8, 24, and 48 weeks
  Changes in HRQoL will be assessed by a questionnaire, which has a total score between 9 to 63. Higher scores are interpreted to a higher quality of life (better outcome).
Changes in the stool microbiome and transcriptome | 8 week
  Stool samples will be collected and after RNA extraction, reverse transcriptase qPCR will be performed. Small RNA sequencing libraries will also be constructed and16S rRNA gene analysis will be conducted.
Safety assessment (Incidence of Treatment-Emergent Adverse Events) | 8 week
  Any adverse events such as Gastrointestinal disorders, Psychiatric disorders, Nervous system disorders, and Immune system disorders will be assessed by the Common Terminology Criteria for Adverse Events Questionnaire.
Changes in the anxiety | 8, 24, and 48 weeks
  Changes in anxiety will be assessed by Beck questionnaire, which has a total score between 0 to 63. Higher scores are interpreted to higher anxiety (worse outcome).
Changes in the metabolomic profile of urine, stool, and saliva | 8 weeks
  Nuclear magnetic resonance will be used for assessment of the metabolomic profile of urine, stool, and saliva